CLINICAL TRIAL: NCT06501157
Title: Establishment of Emergency Surgery Triage and Checklist Management System--A Mixed Method Study
Brief Title: Establishment of Emergency Surgery Triage and Checklist Management System
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: I-24PJ1128
Record Dates: First submitted 2024-06-12; First posted 2024-07-15 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Emergency Surgery; Triage; Checklist; Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- after implementation: Patients undergoing emergency surgery at Peking Union Medical College Hospital after Emergency Surgery Triage and Checklist Management System

SUMMARY:
The goal of this observational study is to develop and test a system for managing emergency surgery patients at Beijing Union Medical College Hospital. The main questions it aims to answer are:

What information is necessary for effective patient triage and handovers between the emergency department, anesthesia, and ICU for surgical patients? How effective and feasible is a standardized handover process in improving patient outcomes and safety?

Participants will:

Be observed and have their handovers documented to identify key information required.

Participate in implementing a new handover checklist and triage system.

Researchers will compare the periods before and after implementing the new system to see if it:

Reduces missed critical information during handovers. Decreases pre-surgery waiting times for critically ill patients. Improves overall patient safety and outcomes, including reducing postoperative complications, mortality rates, length of hospital stay, and medical costs.

DETAILED DESCRIPTION:
The study will be conducted in several phases to establish a comprehensive emergency surgery triage and checklist management system at Beijing Union Medical College Hospital.

Phase 1: Literature Review and Initial Assessment First, a comprehensive review of existing literature and past emergency surgery cases will be conducted to identify common issues and best practices.

Phase 2: Expert Panel and Delphi Process An expert panel consisting of hospital management staff, anesthesiologists, emergency surgeons, ICU intensivists, and ER doctors will be formed. This panel will engage in a Delphi process to discuss and develop a standardized system for managing emergency surgery patients.

Phase 3: System Implementation and Testing

The newly developed system will be implemented and tested. Key metrics to be documented, evaluated, and compared include:

The number of omitted information items during the emergency-anesthesia handover.

Staff satisfaction with the new handover process across the emergency department, general surgery, anesthesia, and ICU.

In-hospital mortality rate after surgery. Postoperative in-hospital complications, classified by Clavien-Dindo grading, and their incidence rate.

Patient waiting times, including time to theatre and time to incision. Duration of the handover process. Incidence of follow-up calls to inquire about additional information after the handover.

Phase 4: Evaluation and Comparison The effectiveness and feasibility of the new system will be evaluated by comparing the collected data before and after its implementation. This comparison will help determine the system's impact on improving patient outcomes, safety, and staff efficiency.

By systematically addressing the critical points of patient handovers and emergency surgery management, this study aims to enhance overall healthcare quality and patient safety in emergency surgical settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for emergency surgery.
* Patients whose condition is critical before surgery, requiring admission to the resuscitation room, emergency observation, or other hospital wards for treatment.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for emergency surgery at Peking Union Medical College Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of omitted information | Outcome will be assessed on the operative day
  The number of omitted information items during the emergency-anesthesia handover.

SECONDARY OUTCOMES:
Patient waiting times, including time to theatre and time to incision. | Outcome will be assessed on the operative day
  Time to Theatre (TTT): This is defined as the duration from when it is determined that the patient needs surgery to the time the patient arrives at the operating theatre. Time to Knife (TTK): This is defined as the duration from when the patient enters the operating theatre to the time the first incision is made.
Feasibility of handover checklist | Outcome will be assessed on the operative day
  Staff satisfaction with the new handover process across the emergency department, general surgery, anesthesia, and ICU. Whether the handover checklist is considered necessary will and feasible will be assessed using a 5 point Likert scale.
In-hospital mortality | From date of admission until discharge, assessed up to 4 weeks
  In-hospital mortality
In-hospital morbidity | From date of admission until discharge, assessed up to 4 weeks
  In-hospital morbidity will be documented and rated using Clavein-Dindo classification system

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No